CLINICAL TRIAL: NCT01897584
Title: Effect of Inverse Ratioventilation on Laparoscopic Low Anterior Resection
Brief Title: Effect Inverse Ratio Ventilation on Arterial Oxygenation and Respiratory Mechanics During lapaLAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gachon University Gil Medical Center (Other)
Responsible Party: Principal Investigator, Youn Yi Jo, Assistant professor, Gachon University Gil Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: GBIRB2013-127; GBIRB2013-127 (Registry Identifier: GIRB)
Record Dates: First submitted 2013-06-26; First posted 2013-07-12 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Colorectal Neoplasms
Keywords: laparoscopy, Trendelenburg Position, ventilation
MeSH Terms: conditions — Colorectal Neoplasms; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Inverse IE (Experimental): in only one group, inspiration to expiration ratio 1:2 to 1:1 will be applied during pneumoperitoneum
  Interventions: Other: inverse IE

INTERVENTIONS:
Other: inverse IE — in only one group changes of I:E ratio would be applied
  Other Names: inverse I:E

SUMMARY:
Changes of inspiration: expiration ration from 1:2 to 1:1 could improve the arterial oxygenation and respiratory mechanics

DETAILED DESCRIPTION:
Inverse ratio ventilation already known as effective to improve the oxygenation and respiratory mechanics in the ARDS patients. Recently, there were report of decrease in airway pressure and improve in respiratory compliance during inverse ration ventilation undergoing one lung ventilation. We hypothesized that changes of inspiration and expiration ratio from 1:2 to 1:1 could improve the arterial oxygenation and respiratory mechanics in the patients who undergoing laparoscopic low anterior resection. However, prolonged inspiratory time might compromise cerebral perfusion pressure due to an elevation in central venous pressure and concomitant reductions in mean arterial pressure.

ELIGIBILITY:
Inclusion Criteria:

* colorectal cancer

Exclusion Criteria:

* obesity (BMI>35), uncontrolled hypertension, coronary artery disease, uncompensated cardiovascular disease, current respiratory disease, open procedure

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2013-07; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
arterial oxygenation (PaO2) | baseline PaO2- 2 hour after pneumoperitoneum
  sampling for arterial blood from arterial cannular will be analyzed 10 min after anesthetic induction, 20 min after pneumoperitoneum, 40 min after pneumoperitoneum and operation end.

SECONDARY OUTCOMES:
cerebral perfusion pressure | immediately before pneumoperitoneum in the Trendelenburg position, every 5 min up to 20 after I:E ratio 1:1
  cerebral perfusion pressure would calculate as mean arterial pressure-central venous pressure from immediately before pneumoperitoneum in the Trendelenburg position, every 5 min up to 20 after I:E ratio 1:1.

CONTACTS AND LOCATIONS:
Overall Officials: Hyun Jeong Kwak, M.D., Ph.D, Study Director — Gachon University Gil Medical Center
Locations (1):
- Kyung Cheon Lee, Incheon, South Korea